CLINICAL TRIAL: NCT06472700
Title: The Feasibility Analysis of Endoscopic Extirpation of Benign Breast Tumors Using Lateral Chest Wall Incision: The Feasibility Analysis of Minimally Invasive Excision for Benign Breast Tumors Via Lateral Chest Wall Approach
Brief Title: Endoscopic Extirpation of Benign Breast Tumors Using a Lateral Chest Wall Incision
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jinghua Zhao, Dr., Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SunYatsenU8H
Record Dates: First submitted 2024-06-15; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Endoscopic Breast Surgery; Benign Breast Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation group
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
1. A new surgical method for breast surgery has been introduced, which involves the removal of benign breast tumors through endoscopic surgery, thereby avoiding noticeable scarring on the breast.
2. The feasibility of this surgery, key technical points, and potential complications have been analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Female breast benign tumor patients
2. Received endoscopic resection of benign breast tumors via a lateral chest wall approach.

Exclusion Criteria:

1. Patients who are unable to comply with follow-up requirements
2. Patients with a history of breast sugery
3. Breast cancer patients

Ages: 14 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population consisted of patients diagnosed with benign breast tumors. The demographic characteristics included:
  Age: Patients aged 14-42 years old Gender: Female Ethnicity: Diverse ethnic backgrounds, primarily Han Chinese
  Inclusion Criteria:
  1. Female breast benign tumor patients
  2. Received endoscopic resection of benign breast tumors via a lateral chest wall approach.
  Exclusion Criteria:
  Patients who are unable to comply with follow-up requirements
  Sample Size:
  A total of 42 patients were included in the study
  Geographical Location:
  Patients were recruited from Sun Yat-sen Memorial Hospital of Sun Yat-sen University
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Cosmetic Outcome After Endoscopic Benign Breast Tumor Resection | 1-3 months post-surgery.
  Through outpatient questionnaires and physician-rated photo evaluations

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China